CLINICAL TRIAL: NCT03750292
Title: Residential Cleaning of Indoor Air to Reduce Acute Exacerbations of COPD (CARE): A Pilot Randomized Crossover Trial
Brief Title: Residential Cleaning of Indoor Air to Protect COPD Patients
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Dan Croft, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 72609
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HEPAirX air filter (Experimental)
  Interventions: Device: HEPAirX air filter
- Control air filter (Placebo Comparator)
  Interventions: Device: control air filter

INTERVENTIONS:
Device: HEPAirX air filter — It is a trademarked, patented (U.S. Patent # 7,802,443), U.S. FDA approved Class II medical re-circulating air cleaner, built by Air Innovations, Inc. (North Syracuse, NY) to provide improved indoor air quality in the bedrooms of asthmatic children. Units to be used in the proposed study have a 99.97% efficient filter for particles 0.3 µm in size. The device provides a clean air delivery rate (CADR) of 9 per hour with 1.8 of them being outdoor air.
  Arms: HEPAirX air filter
Device: control air filter — A placebo mode was added to the HEPAirX to provide only recirculation (without filtration or ventilation using outdoor air) and temperature control of the room air. The placebo filter is made of metal.
  Arms: Control air filter

SUMMARY:
This study looks at whether air cleaning devices put in the bedroom and living room of your home could reduce the irritation of your lungs and body that is caused by indoor air pollution. While participating in this study there will be two, 2 month long study segments (Study Period 1 and Study Period 2) where the air filter units, placed in your living room and bedroom windows, will be turned on at your home.

ELIGIBILITY:
Inclusion Criteria:

* severe COPD (FEV1 < 50%)
* live in Monroe County
* referred for pulmonary rehabilitation
* suffered from an AECOPD in the past year
* have standard sized windows in their bedroom and living room amenable to installation of the HEPAirX® device
* expect to sleep each night of the 4 months (2 months of Period 1, and 2 months of period 2) in either their bedroom or living room for at least 6 hours/night, and not use other air filtering devices during the study

Exclusion Criteria:

* under age 18
* smoking at the time of their prior COPD exacerbation
* current smokers
* those who live with an active smoker
* those with an occupation that has a high pollutant exposure (e.g. professional drivers)
* those who already have a home air filtration device (other than basic furnace filter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Filtration Followed by Placebo: Participants had a HEPAir X air filter in the home for 8 weeks followed by a 3 week washout period and then a placebo period of 8 weeks where the HEPAirX provided only recirculation without filtration or ventilation using outdoor air.
  HEPAirX air filter: It is a trademarked, patented (U.S. Patent # 7,802,443), U.S. FDA approved Class II medical re-circulating air cleaner, built by Air Innovations, Inc. (North Syracuse, NY) to provide improved indoor air quality in the bedrooms of asthmatic children. Units to be used in the proposed study have a 99.97% efficient filter for particles 0.3 µm in size. The device provides a clean air delivery rate (CADR) of 9 per hour with 1.8 of them being outdoor air.
- Placebo Followed by Filtration: Participants had a placebo period of 8 weeks where the HEPAirX provided only recirculation without filtration or ventilation using outdoor airfilter in the home followed by a 3 week washout period and then the HEPAirX air filter for 8 weeks.
  HEPAirX air filter: It is a trademarked, patented (U.S. Patent # 7,802,443), U.S. FDA approved Class II medical re-circulating air cleaner, built by Air Innovations, Inc. (North Syracuse, NY) to provide improved indoor air quality in the bedrooms of asthmatic children. Units to be used in the proposed study have a 99.97% efficient filter for particles 0.3 µm in size. The device provides a clean air delivery rate (CADR) of 9 per hour with 1.8 of them being outdoor air.
Period: First Intervention (Baseline to 8 Weeks)
Arm/Group | Filtration Followed by Placebo | Placebo Followed by Filtration
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Washout (3 Weeks)
Arm/Group | Filtration Followed by Placebo | Placebo Followed by Filtration
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Second Intervention (11 to 19 Weeks)
Arm/Group | Filtration Followed by Placebo | Placebo Followed by Filtration
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.44 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Number of participants with obstructive sleep apnea [Count of Participants; unit: Participants] | 4
Number of participants with Asthma [Count of Participants; unit: Participants] | 1
Number of participants with chronic heart failure [Count of Participants; unit: Participants] | 3
number of participants with diabetes [Count of Participants; unit: Participants] | 2
Number of participants with chronic kidney disease [Count of Participants; unit: Participants] | 2
Number of participants with sinus disease [Count of Participants; unit: Participants] | 2
Number of participants with vitamin D deficiency [Count of Participants; unit: Participants] | 0
Number of participants with a psychiatric condition [Count of Participants; unit: Participants] | 9
Mean smoking pack years [Mean (Standard Deviation); unit: years] | 47.83 (17.59)
Number of participants with COPD symptoms [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in St. George Respiratory Questionnaire
Description: The St. Georges Respiratory Questionnaire (SGRQ) is an established, clinically relevant measure of respiratory symptoms, activity level, and impacts on daily life, and is a measure of functional status regularly used and validated in COPD patient populations. The questionnaire is a fixed format 50 item survey completed by the study subject asking questions in three parts: 1) levels of symptomatology including frequency of wheezing, cough, sputum production, and breathlessness, including the duration of episodes of wheeze and breathlessness, 2) physical activities that may be caused or are limited by breathlessness, and 3) impacts of these symptoms. It is a self-assessment of respiratory symptoms and functional status, and provides a quantification of the impacts of airflow limitation on health and well-being. The scores range from 0 to 100 with higher number indicating worse outcomes.
Time Frame: baseline to 8 weeks
Population: Baseline data was not collected on one subject in the HEPAirX air filter arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 4 | 4
score on a scale | -12.5 (20.00) | -0.45 (7.47)

2. Primary Outcome: Mean Change in St. George Respiratory Questionnaire
Description: as for outcome 1
Time Frame: 11 weeks to 19 weeks
Population: Data was not collected on one subject in the HEPAirX air filter arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 4 | 4
score on a scale | 9.65 (13.4) | 1.68 (1.88)

3. Primary Outcome: Mean Change in St. George Respiratory Questionnaire
Description: as for outcome 1
Time Frame: week 19 to week 31
Population: Data was collected on only three patients made it to week 31, two in the placebo arm and one in the filter arm. Therefore an measure of dispersion/precision could not be provided.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 1 | 2
score on a scale | 21.3 [21.3 to 21.3] | 1.14 [-6.28 to 8.55]

4. Primary Outcome: Mean Change in Daily Steps
Description: Steps will be measured using a Fitbit step counter.
Time Frame: week 0 to week 8
Population: Data was not collected on one subject in the HEPAirX air filter arm.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 4 | 4
steps per day | 6.43 (111.47) | -16.57 (23.98)

5. Primary Outcome: Mean Change in Daily Step
Description: Steps will be measured using a Fitbit step counter.
Time Frame: 11 weeks to 19 weeks
Population: Data was not collected on one subject in the HEPAirX air filter arm.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 4 | 4
steps per day | 39.41 (78.66) | -3.85 (100.67)

6. Secondary Outcome: Mean Plasma C-reactive Protein Level
Description: Plasma C-reactive protein (CRP) is a measure of systemic inflammation, and is an acute phase protein known to increase in the hours and days following an inflammatory stimulus. C-reactive protein will be measured in plasma obtained from whole blood using standard procedures.
Time Frame: week 0 to week 19
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 9 | 9
mg/L | 9.75 (13.84) | 5.9 (7.72)

7. Secondary Outcome: Mean Number of Outpatient and Inpatient Visits for Chronic Obstructive Pulmonary Disorder Exacerbations
Description: The number of exacerbations will be measured using retrospective review of Patient charts.
Time Frame: baseline to week 31
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 5 | 4
visits | 1 (0) | 1 (0)

8. Secondary Outcome: Mean Number of Outpatient and Inpatient Visit for Chronic Obstructive Pulmonary Disorder Exacerbations
Description: The number of exacerbations will be measured using patient report
Time Frame: baseline to week 31
Population: Data was not collected for this outcome measure.
Arm/Group | HEPAirX Air Filter | Control Air Filter
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 weeks
Arm/Group | HEPAirX Air Filter | Control Air Filter
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03750292/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT03750292/ICF_002.pdf